CLINICAL TRIAL: NCT03618472
Title: Effect of Metformin for Deceasing Proliferative Marker in Endometrial Cancer Cells : a Randomized Double Blind Placebo-controlled Trial
Brief Title: Comparison of the Effectiveness Metformin for Deceasing Proliferative Marker in Endometrial Cancer Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rjmetformin
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2018-10

CONDITIONS: Metformin; CA Endometrium
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- metformin (Experimental): The participant will be eat metformin 850 mg 1 tab daily,4 weeks prior to hysterectomy
  Interventions: Drug: Metformin Hydrochloride 850 MG
- placebo (Placebo Comparator): The participant will be eat placebo (same shape, size, color)1 tab daily ,4 weeks prior to hysterectomy
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Metformin Hydrochloride 850 MG — Regular strength metformin (850 mg/tab)
  Other Names: if any
  Arms: metformin
Drug: Placebo Oral Tablet — Starch based placebo manufatured to mimic Metformin 850 mg
  Other Names: if any
  Arms: placebo

SUMMARY:
Comparison of the effectiveness metformin versus placebo for deceasing proliferative marker Ki-67 expression in endometrial tumours when given for 4 weeks before hysterectomy in endometrial cancer cells.

DETAILED DESCRIPTION:
Endometrial cancer is one of the most common gynecological cancers. Preclinical studies in endometrial cancer (EC) show that metformin reduces cellular proliferation by PI3K-AKT-mTOR inhibition. The investigators tested the hypothesis that short-term presurgical metformin reduces cellular proliferation in endometrial cancer. However, no good quality of evidence base supports the effectiveness of metformin for deceasing proliferative marker in endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women with endometrial cancer who undergoing complete surgical staging and agrees to participate in this study

Exclusion Criteria:

* Women without diabetes type 1 and 2
* Women who have allergy Biguanide
* Women who have hypoglycemic medication
* Women who have GFR <45 ml/min/1.73 m2
* Women who have evidence of stage 3 or 4 of endometrial cancer

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Change of Ki-67 expression in endometrial tumor | 4 weeks
  metformin administration reduced Ki-67 expression in endometrial tumor when given for 4 weeks before hysterectomy.

SECONDARY OUTCOMES:
Change of grade in endometrial tumor | 4 weeks
  metformin administration reduced grade in endometrial tumor when given for 4 weeks before hysterectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Bangkok, Thailand